CLINICAL TRIAL: NCT06530953
Title: Comparing Two Linkage-to-Care Models for Latinx Immigrant Patients : A Pilot Comparative Clinical Effectiveness Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Ann Cheney, Associate Professor, University of California, Riverside
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 30382
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigator/ Community Health Worker (Active Comparator): The community health worker will contact the participant two days after their initial clinic visit. They will call the participant to offer support and counseling on accessing their follow-up visits with local healthcare system. Additionally, the PN will call 1 day prior to the scheduled appointment to offer support and information to the patient followed by a reminder text the morning of the appointment.
  Interventions: Behavioral: Patient Navigator Model
- Patient Navigator/Clinic Staff (Active Comparator): Clinic staff will contact the participant two days after their initial clinic visit. They will call the participant to offer support and counseling on accessing their follow-up visits with local healthcare system. Additionally, the clinic staff will call 1 day prior to the scheduled appointment to offer support and information to the patient followed by a reminder text the morning of the appointment.
  Interventions: Behavioral: Patient Navigator Model

INTERVENTIONS:
Behavioral: Patient Navigator Model — The patient navigator model is an evidence-based intervention to improve access to healthcare services.

SUMMARY:
The goal of this randomized clinical comparative effectiveness trail is to compare the effects of patient navigator models on follow-up care in Latinx and Indigenous Mexican immigrant patient populations. The main question[s] it aims to answer [is/are]:

* Participants randomized to PN-CHW compared to the PN-CS model will be more likely to follow through with follow-up care referrals
* Trust will be a driving factor as to why PN-CHW will be a more effective intervention for the patient population.

Researchers will compare patients in a patient navigator community health worker (PN-CHW) intervention to those in a patient navigator clinical staff (PN-CS) intervention to see which model of linkage to care is more effective for follow-up care in the patient population.

Participants will be asked to:

* Complete a baseline survey about healthcare access
* Receive calls and text messages from either a CHW or clinical staff
* Complete a follow up survey

DETAILED DESCRIPTION:
The research project will be conducted at a free clinic that serves a primarily Spanish-speaking Latinx patient population in the Inland Southern California region. Patients in this study will be randomized to one of two intervention arms: Arm 1: PN model delivered by CHWs/promotoras and Arm 2: PN model delivered by clinic staff. CHWs who live in the region and work at the free clinic will deliver the PN model for Arm 1 participants. CHWs have a detailed knowledge of local health resources, as well as lived experience of the barriers patients in their community face when accessing healthcare services. Medical students who are volunteer clinic staff will deliver the PN model for Arm 2 participants. Medical students are the doctors in training who provide primary care services to patients at the CVFC under the supervision of well-established physicians. Baseline data and follow-up data at 12 weeks will be collected along with qualitative interviews with patients in both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1) live in the Coachella Valley, 2) 18 or older, 3) household income less than or equal to or below 200% of federal poverty guidelines, 4) do not currently have health insurance, and 5) have access to a telephone.

Exclusion Criteria:

* Do not speak English, Spanish or Purépecha (an indigenous dialect spoken among the Purépecha of Mexico).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Follow up care | 12 weeks post randomization
  Follow up care for referred healthcare need

SECONDARY OUTCOMES:
Trust in physicians | 12 weeks post randomization
  Trust in physicians measured by 10-item physician trust Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Cheney, PhD, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request to the study principal investigator.
Supporting Information: CSR
Time Frame: De-identified data will be available after the completion of main analysis and scientific dissemination.
Access Criteria: Interested parties should contact the principal investigator at ann.cheney@medsch.ucr.edu